CLINICAL TRIAL: NCT01507415
Title: Do the SPPB and 4-metre Gait Speed Predict Hospital Readmission in Patients Hospitalised for Acute Exacerbation if COPD?
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government); The Hillingdon Hospitals NHS Foundation Trust (Other Government); West Hertfordshire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2011LF015H
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive; Bronchitis, Chronic; Pulmonary Emphysema; Disease Progression
Keywords: Cohort Studies; Longitudinal Studies; Patient Readmission; Hospitalization; Disability Evaluation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive; Bronchitis, Chronic; Pulmonary Emphysema; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma and serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exacerbation: Patients with Chronic Obstructive Pulmonary Disease (COPD)

SUMMARY:
This study aims to evaluate simple tests of physical function in hospitalised patients with chronic obstructive pulmonary disease (COPD) and to assess whether they can predict future hospital readmission. The Short Physical Performance Battery (SPPB) is a simple test of standing balance, usual walking speed (4-metre gait speed) and ability to stand from a chair, which reflects global physical functioning and frailty.

We hypothesise that the SPPB or 4-metre gait speed can predict future hospital readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission with an exacerbation of COPD
* Must have capacity to consent
* Able to walk

Exclusion Criteria:

* Co-morbibities that limit walking ability
* Co-morbidities that make walking unsafe

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient hospitalised with an acute exacerbation of COPD. Cohorts will be recruited from local District General Hospitals with Acute Admissions Units and Accident & Emergency Departments.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Hospital readmission rate | 3 months

SECONDARY OUTCOMES:
Hospital readmission rate | 12 months
Time to first hospital readmission | 12 months
Hospital Bed days | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, MRCP PhD, Principal Investigator — NIHR Respiratory Biomedical Research Unit, Royal Brompton & Harefield NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Hillingdon Hospital, Uxbridge
  - Watford General Hospital, Watford

REFERENCES:
- [Background] Volpato S, Cavalieri M, Sioulis F, Guerra G, Maraldi C, Zuliani G, Fellin R, Guralnik JM. Predictive value of the Short Physical Performance Battery following hospitalization in older patients. J Gerontol A Biol Sci Med Sci. 2011 Jan;66(1):89-96. doi: 10.1093/gerona/glq167. Epub 2010 Sep 22. PMID 20861145
- [Derived] Nolan CM, Kon SSC, Patel S, Jones SE, Barker RE, Polkey MI, Maddocks M, Man WD. Gait speed and pedestrian crossings in COPD. Thorax. 2018 Feb;73(2):191-192. doi: 10.1136/thoraxjnl-2017-210173. Epub 2017 May 5. PMID 28476882
- [Derived] Kon SS, Jones SE, Schofield SJ, Banya W, Dickson MJ, Canavan JL, Nolan CM, Haselden BM, Polkey MI, Cullinan P, Man WD. Gait speed and readmission following hospitalisation for acute exacerbations of COPD: a prospective study. Thorax. 2015 Dec;70(12):1131-7. doi: 10.1136/thoraxjnl-2015-207046. Epub 2015 Aug 17. PMID 26283709